CLINICAL TRIAL: NCT04560218
Title: Sublingual Versus Intrauterine MISOPROSTOL in Addition to Oxytocin Infusion for Prevention of Post-cesarean Hemorrhage in High Risk Pregnant Women: A Double-blind Randomized Placebo Controlled Trial
Brief Title: Sublingual vs Intrauterine MISOPROSTOL Plus Oxytocin Infusion for Prevention of Post-cesarean Hemorrhage in High Risk Pregnant Women: A Double-blind Placebo RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 122/2563
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-07

CONDITIONS: To Compare Efficacy Intrauterine vs Sublingual MISOPROSTOL in Addition to Oxytocin in Reducing Blood Loss of Post-cesarean Section in High Risk Women
Keywords: Postpartum hemorrhage, Cesarean section, Sublingual Misoprostol, Intrauterine Misoprostol
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Uterotonic agents group A (Experimental): Misoprostol sublingually 2 tab (400 mcg) + Oxytocin 20 IU Intravenous + Placebo Intrauterine 2 tab
  Interventions: Drug: sublingual Misoprostol
- Uterotonic agents group B (Experimental): Misoprostol Intrauterine 2 tab (400 mcg) + Oxytocin 20 IU Intravenous + Placebo sublingually 2 tab
  Interventions: Drug: Intrauterine Misoprostol
- Uterotonic agents group C (No Intervention): Oxytocin 20 IU Intravenous + Placebo Intrauterine 2 tab + Placebo sublingually 2 tab

INTERVENTIONS:
Drug: sublingual Misoprostol — apply drug by Anesthesiologist
  Arms: Uterotonic agents group A
Drug: Intrauterine Misoprostol — apply drug by surgeon at uterine cornu
  Arms: Uterotonic agents group B

SUMMARY:
Research Objective:

Primary outcome

-To compare efficacy Intrauterine vs Sublingual MISOPROSTOL in addition to Oxytocin in reducing blood loss of post-cesarean section in high risk women

Secondary outcome

-To study Hemoglobin/Hematocrit change, need of uterotonic agents, need of blood transfusion, adverse drug event of Intrauterine vs Sublingual Misoprostol plus Oxytocin compare to Oxytocin alone

Hypothesis:

-Intrauterine MISOPROSTOL plus Oxytocin is not inferior to Sublingual MISOPROSTOL plus Oxytocin in reducing blood loss of post-cesarean section in high risk women

DETAILED DESCRIPTION:
Research Design: Double-blind Randomized Placebo Controlled Trial

Subject: Singleton pregnancy GA 34 wk or more with high risk for postpartum hemorrhage undergo cesarean section with spinal anesthesia in Rajavithi Hospital

Allocated to 3 groups

* group1: Misoprostol sublingually 2 tab (400 mcg) + Oxytocin 20 IU Intravenous + Placebo Intrauterine 2 tab
* group2: Misoprostol Intrauterine 2 tab (400 mcg) + Oxytocin 20 IU Intravenous + Placebo sublingually 2 tab
* group3: Oxytocin 20 IU Intravenous + Placebo Intrauterine 2 tab + Placebo sublingually 2 tab

ELIGIBILITY:
Inclusion Criteria:

* ≥35 ปี
* Previous PPH
* Morbid obesity
* Fetal macrosomia
* Polyhydramnios
* Induction/Augmentation of Labour
* Prolonged Labour
* Grand multiparity
* Preeclampsia
* Myoma Uteri

Exclusion Criteria:

* Asthma
* Maternal fever/ Tripple I can't excluded
* coagulopathy
* Placenta previa/ adherens/ abruptio placenta
* Allergy to Prostaglandins/Oxytocin

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 135 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Blood loss | operation time
  total blood loss estimated by Anesthesiologist team

SECONDARY OUTCOMES:
Hemoglobin/Hematocrit change | until 24 hours post-operation
  compare before/after operation
need of uterotonic agents | until 24 hours post-operation
  number of uterotonic agents need and type of drug
need of blood transfusion | until 24 hours post-operation
  number of blood transfusion need
adverse drug event | until 24 hours post-operation
  adverse drug event of Misoprostol and Oxytocin

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi hospital, Bangkok, Thailand